CLINICAL TRIAL: NCT03838133
Title: A Phase 2, Randomized, Double-blind, Comparator- and Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of TLC590 for Postsurgical Pain Management Following Bunionectomy
Brief Title: A Study to Evaluate Safety, PK, Efficacy of TLC590 for Postsurgical Pain Management Following Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: TLC590A1002
Record Dates: First submitted 2019-02-11; First posted 2019-02-12 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus | interventions — Ropivacaine; Saline Solution; Sodium Chloride; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- TLC590 dose 1 (152 mg) (Experimental): TLC590 (Ropivacaine Liposome Injectable Suspension) is a sustained-release liposome formulation of ropivacaine, white aqueous suspension with ropivacaine concentration at approximately 19 mg/mL.
  Interventions: Drug: TLC590
- TLC590 dose 2 (190 mg) (Experimental): TLC590 (Ropivacaine Liposome Injectable Suspension) is a sustained-release liposome formulation of ropivacaine, white aqueous suspension with ropivacaine concentration at approximately 19 mg/mL.
  Interventions: Drug: TLC590
- TLC590 dose 3 (228 mg) (Experimental): TLC590 (Ropivacaine Liposome Injectable Suspension) is a sustained-release liposome formulation of ropivacaine, white aqueous suspension with ropivacaine concentration at approximately 19 mg/mL.
  Interventions: Drug: TLC590
- Naropin® (Active Comparator): Naronpin injection contains ropivacaine HCl 50 mg (0.5%, 10 mL)
  Interventions: Drug: Naropin®
- Placebo (Placebo Comparator): Normal Saline (0.9% sodium chloride, 10 mL)
  Interventions: Drug: Normal Saline
- Bupivacaine (Active Comparator): Bupivacaine HCl 50 mg (0.5%, 10 mL)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: TLC590 — TLC590, a sustained-release formulation of the local anesthetics with lipid-based excipients
  Other Names: TLC590 (Ropivacaine Liposome Injectable Suspension)
  Arms: TLC590 dose 1 (152 mg); TLC590 dose 2 (190 mg); TLC590 dose 3 (228 mg)
Drug: Naropin® — Local infiltration of Naropin to produce anesthesia for surgery and analgesia in postoperative pain management. 50 mg (0.5%, 10 mL)
  Other Names: Naropin, 0.5% Injectable Solution
  Arms: Naropin®
Drug: Normal Saline — Normal Saline (0.9% sodium chloride, 10ml)
  Other Names: Saline
  Arms: Placebo
Drug: Bupivacaine — Bupivacaine 50 mg (0.5%, 10 mL)
  Arms: Bupivacaine

SUMMARY:
This is a Phase 2, randomized, double-blind, 2-part comparator- and placebo-controlled study to evaluate the safety, PK, and efficacy of TLC590 via a single infiltrative local administration in adult subjects following bunionectomy.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, 2-part comparator- and placebo-controlled study to evaluate the safety, PK, and efficacy of TLC590 via a single infiltrative local administration in adult subjects following bunionectomy.

The primary objective of this study is to evaluate the analgesic efficacy of TLC590 for post-surgical pain management in subjects following bunionectomy.

The secondary objectives of this study are:

* To evaluate the pharmacokinetic (PK) profile and dose-exposure relationship of TLC590, as well as the bioavailability as compared with Naropin®.
* To evaluate the safety and tolerability of TLC590 for post-surgical pain management in subjects following bunionectomy.
* To evaluate the exposure-response relationship between PK parameters and pain intensity.

The study will be divided into two parts:

Part 1: Blinded Pharmacokinetics of TLC590 and Naropin®. Approximately 48 subjects will be randomized to treatments.

Part 2: Efficacy and Safety of TLC590 versus bupivacaine and Placebo. Part 2 of the study will randomize approximately 150 evaluable subjects who meet all entry criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Male or female between 18 and 65 years of age.
3. Body mass index ≤ 35 kg/m2.
4. Mild to moderate hallux valgus deformity.
5. Scheduled to undergo a primary, unilateral first metatarsal bunionectomy repair under local anesthesia.
6. American Society of Anesthesiology Physical Status Classification of 1 or 2 at screening.
7. Female subjects are eligible only if all of the following apply:

   * Not pregnant;
   * Not lactating;
   * Not planning to become pregnant during the study;
   * Commits to the use of an acceptable form of birth control for the duration of the study and for 42 days from administration of study drug.
8. Male subjects must be surgically sterile (biologically or surgically) or commit to the use of a reliable method of birth control, for the duration of the study until at least 1 week after the administration of study medication.

Exclusion Criteria:

1. Clinically significant abnormal clinical laboratory test value.
2. Evidence of a clinically significant 12-lead ECG abnormality.
3. History or evidence of orthostatic hypotension, syncope or other syncopal attacks.
4. History or clinical manifestations of significant renal, hepatic, gastrointestinal, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study.
5. A history of seizure disorder or currently taking anticonvulsants.
6. History of hypersensitivity to ropivacaine, any other amide-type local anesthetic, propofol, lidocaine, midazolam, acetaminophen, naproxen, morphine or oxycodone (or other opioids).
7. Concurrent painful physical condition that may confound post-operative pain assessments.
8. Persistent or recurrent nausea and/or vomiting due to other etiologies.
9. History of severe or refractory post-operative nausea or vomiting (PONV) deemed clinically significant.
10. History of alcohol abuse or prescription/illicit drug abuse within 2 years.
11. Current evidence of alcohol abuse within 6 months.
12. Received opioid therapy for longer than 4 days per week within 2 months or opioid use within 2 weeks.
13. Use of concurrent therapy that could interfere with the evaluation of efficacy or safety.
14. Unable to discontinue medications that have not been at a stable dose for at least 14 days prior to the study surgical procedure, within 5 half-lives of the specific prior medication.
15. Use of any of the following medications within 5 half-lives or as specified prior to the study surgical procedure:

    * Low-dose aspirin therapy for cardiovascular protection
    * Class III antiarrhythmic drugs
    * Strong CYP1A2 inhibitors
    * CYP1A2 substrates
    * Strong CYP3A4 inhibitors
    * Corticosteroids, either systemically, inhaled either intranasally or orally, or by intra-articular injection, or NSAIDs within 14 days
    * Any investigational product within 30 days.
16. Positive results on the urine drug screen or alcohol breath test indicative of illicit drug or alcohol abuse.
17. History or positive test results for HIV; active Hepatitis B or C.
18. Contralateral foot bunionectomy in the last 3 months or have collateral procedures.
19. Malignancy in the last 2 years, with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
20. History of rheumatoid disease, Type 1 or Type 2 diabetes or peripheral circulatory disorders.
21. Documented sleep apnea or are on home continuous positive airway pressure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
AUC of numerical pain rating scale | 0-24 hours, 0-72 hours
  AUC of numerical pain rating scale (NPRS-R) following bunionectomy surgery

SECONDARY OUTCOMES:
PK Cmax | 0-168 hours
  Maximum blood concentration (Cmax)
PK Tmax | 0-168 hours
  Time to reach maximum blood concentration (Tmax)
PK t½ | 0-168 hours
  Terminal elimination half-life (t½)
PK AUC | 0-24, 0-48 , 0-72, 0-96 hours
  Area under the blood concentration-time curve (AUC)
Number of treatment emergent adverse event (TEAE) | Screening through Day 43
  Number of treatment emergent adverse event (TEAE) occurred in the study
Electrocardiogram (RR interval, QRS duration, QT duration, PR duration, QTcF interval) | Screening through Day 43
  The 12-lead electrocardiogram (ECG) result will be assessed including RR interval, QRS duration, QT duration, PR duration, and QTcF interval
Wound assessment by Numerical Pain Rating Scale (NPRS) | Day 1 through Day 43
  The surgical site will be examined by the investigator using a 5-point numerical pain rating scale as follows:
  1. Normal healing
  2. Bruising, erythema, edema
  3. Clear or hemoserous drainage
  4. Evidence of cellulitis such as heat, spreading erythema, purulent discharge
  5. Tissue breakdown, wound dehiscence, hematoma requiring aspiration
AUC of NPRS-R (0-10) | 0-36, 0-48, 0-72, 0-96, 0-120,24-48, 48-72, 72-96, 96-120, and 120-168 hours
  AUC of NPRS-R (0-10)
Proportion of pain-free (NPRS-R of 0 or 1) subjects | at 12, 24, 36, 48, 72, 96, 120, and 168 hours
  Proportion of pain-free (NPRS-R of 0 or 1) subjects
Proportion of subjects who used no rescue opioid analgesic | through 12, 24, 36, 48, 72, 96, 120, and 168 hours
  Proportion of subjects who used no rescue opioid analgesic
Time to the first postoperative use of rescue opioid analgesics | Day 1 to Day 43
  Time to the first postoperative use of rescue opioid analgesics
Total postoperative consumption of rescue opioid analgesics used | through 24, 36, 48, 60, 72, 96, 120, and 168 hours
  Total postoperative consumption of rescue opioid analgesics used

CONTACTS AND LOCATIONS:
Overall Officials: Carl Brown, PhD, Study Director — Taiwan Liposome Company
Locations (5):
- United States (5):
  - Arizona Research Center, Phoenix, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Chesapeake Research Group, Pasadena, Maryland
  - Endeavor Clinical Trials, San Antonio, Texas
  - JBR clinical research, Draper, Utah

IPD SHARING:
Plan to Share IPD: No